CLINICAL TRIAL: NCT04693195
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Evaluate the Efficacy, Safety, and Tolerability of BLU-5937 for the Treatment of Chronic Pruritus in Adult Subjects With Atopic Dermatitis
Brief Title: A Multiple-Dose Study of BLU-5937 in Chronic Pruritus Associated With Atopic Dermatitis
Acronym: BLUEPRINT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-PR-5937-01
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Chronic Pruritus; Atopic Dermatitis
Keywords: BLU-5937; Chronic Pruritus; Atopic Dermatitis; P2X3 receptor antagonist
MeSH Terms: conditions — Dermatitis, Atopic | interventions — BLU-5937

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BLU-5937 oral tablet (Experimental): Eligible participants will receive BLU-5937 twice a day (BID) orally for 4 weeks.
  Interventions: Drug: BLU-5937
- Placebo oral tablet (Placebo Comparator): Eligible participants will receive matching Placebo BID orally for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BLU-5937 — Oral administration of BLU-5937 tablets
  Arms: BLU-5937 oral tablet
Drug: Placebo — Oral administration of matching placebo for BLU-5937 tablets
  Arms: Placebo oral tablet

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel design study of BLU-5937 for the treatment of chronic pruritus in adult subjects with atopic dermatitis (AD).

DETAILED DESCRIPTION:
The study will consist of a 37-day Screening period (including a 7-day Run-In period), a 4-week Treatment period followed by a Follow-Up visit approximately 2 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate and is capable of giving informed consent
* Clinically confirmed diagnosis of active AD with at least a 6-month history of AD
* Chronic pruritus related to AD for at least 3 months
* Moderate to severe itch associated with mild to moderate AD
* Female of childbearing potential must agree to use a highly effective contraceptive method during the study and until at least 4 weeks after the last study drug administration

Exclusion Criteria:

* History of skin disease or presence of skin condition that would interfere with the study assessments
* Clearly defined etiology for pruritus other than AD, including but not limited to: urticaria, psoriasis, or other non-atopic dermatologic conditions, hepatic or renal disease, psychogenic pruritus, drug reaction, uncontrolled hyperthyroidism, and infection
* Presence of any acute skin condition other than AD which may risk inducing a pruritus flare/worsening during the course of the study, including but not limited to: impetigo, active herpes simplex infection, or allergic contact dermatitis
* Subject is >65 years of age and has developed pruritus at age of ≥50 years
* History of cancer or lymphoproliferative disease within 5 years with the exception of successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix
* Known history of, or active, parasitic infection, including skin parasites such as scabies within 12 months prior to Screening
* Known history of chronic infectious disease (e.g. hepatitis B, hepatitis C, or human immunodeficiency virus [HIV])
* Known history of clinically significant drug or alcohol abuse in the last year
* Previous participation in a BLU-5937 trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weekly mean Worst Itch Numeric Rating Scale (WI-NRS) score | Week 4
  Assessed by Worst Itch Numeric Rating Scale [WI-NRS]
  The WI-NRS is a single item questionnaire assessing the patient-reported severity of itch at its most intense during the previous 24-hour period on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'the worst itch imaginable'. Higher scores indicate worse severity.

SECONDARY OUTCOMES:
Proportion of subjects achieving at least 4-point improvement from baseline in weekly mean Worst Itch Numeric Rating Scale (WI-NRS) score | Week 4
  Assessed by Worst Itch Numeric Rating Scale [WI-NRS]
  The WI-NRS is a single item questionnaire assessing the patient-reported severity of itch at its most intense during the previous 24-hour period on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'the worst itch imaginable'. Higher scores indicate worse severity.
Change from baseline in Average Itch Numeric Rating Scale (AI-NRS) score | Week 4
  Assessed by Average Itch Numeric Rating Scale [AI-NRS]
  The AI-NRS is a single item questionnaire assessing the patient-reported severity of itch overall (on average) during the previous 24-hour period on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'the worst itch imaginable'. Higher scores indicate worse severity.
Change from baseline in Itching Quality of Life Survey (ItchyQOL) | Week 4
  Assessed by Itching Quality of Life Survey [ItchyQOL]
  The ItchyQOL is a 22-item questionnaire assessing the pruritus-specific disease burden on 3 domains: symptoms, functions and emotions. The responses to the frequency items are scored on a 1 (never) to 5 (all the time) scale. The recall period in ItchyQoL is the past week. Higher scores indicate a more adverse impact on quality of life.
Proportion of subjects in each category of the Patient Global Impression of Change (PGIC) questionnaire | Week 4
  Assessed by Patient Global Impression of Change [PGIC]
  The PGIC consists of 1 self-administered item that assesses the subject's impression of change in the severity of pruritus using a 7-point scale from 1 (very much improved) to 7 (very much worse). Higher scores indicate a worsening of the severity.

CONTACTS AND LOCATIONS:
Locations (33):
- United States (28):
  - Bellus Health Investigational Site #28, Phoenix, Arizona
  - Bellus Health Investigational Site #10, Scottsdale, Arizona
  - Bellus Health Investigational Site #23, Beverly Hills, California
  - Bellus Health Investigational Site #33, Encinitas, California
  - Bellus Health Investigational Site #27, Fountain Valley, California
  - Bellus Health Investigational Site #35, San Diego, California
  - Bellus Health Investigational Site #15, Hialeah, Florida
  - Bellus Health Investigational Site #32, Margate, Florida
  - Bellus Health Investigational Site #16, Miami, Florida
  - Bellus Health Investigational Site #19, Miami, Florida
  - Bellus Health Investigational Site #17, Sweetwater, Florida
  - Bellus Health Investigational Site #24, Savannah, Georgia
  - Bellus Health Investigational Site #13, Owensboro, Kentucky
  - Bellus Health Investigational Site #38, Baton Rouge, Louisiana
  - Bellus Health Investigational Site #45, Covington, Louisiana
  - Bellus Health Investigational Site #18, New Orleans, Louisiana
  - Bellus Health Investigational Site #36, Minneapolis, Minnesota
  - Bellus Health Investigational Site #22, Portsmouth, New Hampshire
  - Bellus Health Investigational Site #34, New York, New York
  - Bellus Health Investigational Site #14, High Point, North Carolina
  - Bellus Health Investigational Site #29, Norman, Oklahoma
  - Bellus Health Investigational Site #37, Newtown Square, Pennsylvania
  - Bellus Health Investigational Site #41, Rapid City, South Dakota
  - Bellus Health Investigational Site #12, Austin, Texas
  - Bellus Health Investigational Site #31, College Station, Texas
  - Bellus Health Investigational Site #40, San Antonio, Texas
  - Bellus Health Investigational Site #11, San Antonio, Texas
  - Bellus Health Investigational Site #25, Seattle, Washington
- Canada (5):
  - Bellus Health Investigational Site #44, Chicoutimi, Quebec
  - Bellus Health Investigational Site #20, Montreal, Quebec
  - Bellus Health Investigational Site #43, Québec, Quebec
  - Bellus Health Investigational Site #39, Québec, Quebec
  - Bellus Health Investigational Site #42, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No